CLINICAL TRIAL: NCT03460639
Title: Administration of Low-level Laser on Muscles of Mastication Following the Induction of Initial Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Greice de Brito Bitencourt, Principal investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 919822905; 290582 (Other: uninove)
Record Dates: First submitted 2017-12-05; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Muscle Fatigue
Keywords: Masseter muscle; initial fatigue; low-level laser

STUDY DESIGN:
Intervention Model Description: Tiredness will be induced by isometric contraction occlusion time. Patients will be evaluated in two stages. The first moment will be maximum occlusion in all patients in order to be able to measure the individual time for fatigue of the masseter muscle (evaluation by electromyography). The second will have the application of the laser in a group (at the wavelength of 780nm, 134 J / cm2, power of 50 mW irradiance of 1.675 W / cm2, for 80 seconds per point in 3 points in the masseter muscle and one in the temporal muscle on each side); simulation of the application (placebo-psychic factor), control (without application); after this first moment, we will have maximum occlusion in all the patients in order to be able to measure the individual time for fatigue (evaluation by electromyography).
Who Masked: Participant
Masking Description: In the sham group, the laser will be switched off and a recording of the emission sounds will be used to give the volunteer the auditory sensation of laser therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active laser (Active Comparator): Three points on the masseter muscle (upper, middle and lower portions) and one point on the anterior temporal on each side of the face will be irradiated with a wavelength of 780 nm, radiant exposure of 134 J/cm2, power of 50 mW and irradiance of 1.675 W/cm2 for 80 seconds per point, resulting in an energy of 4 J per point and total energy of 32 J per volunteer.20,21 Point application will be performed with a conventional tip in contact with the skin (beam spot: 0.04 cm2).
  Interventions: Radiation: Active laser
- Sham laser (Sham Comparator): The same procedures will be performed in the sham group, but the device will be switched off and a recording of the emission sounds will be used to give the volunteer the auditory sensation of laser therapy.
  Interventions: Radiation: Sham laser
- Control group (Other): In this group, no treatment will be done, we will only induce fatigue, for evaluation.
  Interventions: Diagnostic Test: Control group

INTERVENTIONS:
Radiation: Active laser — Three points on the masseter muscle (upper, middle and lower portions) and one point on the anterior temporal on each side of the face will be irradiated with a wavelength of 780 nm, radiant exposure of 134 J/cm2, power of 50 mW and irradiance of 1.675 W/cm2 for 80 seconds per point, resulting in an energy of 4 J per point and total energy of 32 J per volunteer.20,21 Point application will be performed with a conventional tip in contact with the skin (beam spot: 0.04 cm2).
  Arms: Active laser
Radiation: Sham laser — The same procedures will be performed in the sham group, but the device will be switched off and a recording of the emission sounds will be used to give the volunteer the auditory sensation of laser therapy.
  Arms: Sham laser
Diagnostic Test: Control group — In this group, we will only induce fatigue.
  Arms: Control group

SUMMARY:
Orofacial pain encompasses painful conditions, such as temporomandibular disorder. Multidisciplinary health teams seek to control such musculoskeletal disorders to improve the quality and functional capacity of the muscles of mastication. The aim of the proposed study is to evaluate the effect of low-level laser therapy as a form of treatment for the prevention of initial fatigue of the muscles of mastication (masseter and anterior temporal muscles) as well as the recovery of these muscles after induced exhaustion (caused by isometric contraction) in young adults. The participants will be 78 (n obtained from calculation of the sample size with p < 0.05) healthy male and female volunteers between 18 and 34 years of age. The volunteers will be randomly allocated to a laser group (n = 26), sham group (n = 26) and control group (n = 26). All participants will be submitted to a clinical evaluation to record mandibular movements, bite force, muscle sensitivity to palpation and initial muscle fatigue. Initial fatigue will be induced by isometric contraction of the jaws. Maximum voluntary contraction will be performed to record the time until initial exhaustion of the masseter muscle (determined by electromyography). The groups will then be submitted to the interventions: 1) active laser therapy (wavelength: 780 nm; fluence: 134 J/cm2; power: 50 mW; irradiance: 1.675 W/cm2; exposure time: 80 seconds per point) on three points of the masseter and one point on the anterior temporal muscles on each side, 2) sham laser (placebo effect) or 3) no intervention (control). Maximum voluntary contraction will be performed again after the interventions to record the time until initial exhaustion of the masseter muscle (determined by electromyography). Differences in individual time until exhaustion between the pre-intervention and post-intervention evaluations will be measured to determine the effect of low-level laser therapy.

ELIGIBILITY:
Inclusion Criteria:

* will be included in this study young people in the age range between 18-34 years, without diagnosis of temporomandibular disorder (TMD) and with the signed free informed consent term.

Exclusion Criteria:

* will be excluded from the study individuals who are in orthodontic or orthopedic treatment of the jaw, psychological and / or physiotherapy. Also excluded are those who are taking anti-inflammatory drugs and anti-inflammatory drugs and occlusal plaques.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change of the masseter muscle strength determined by electromyography before and after treatment | Before and immediately after treatment
  MVC (clenching the teeth in maximum intercuspation) will be performed to record the time until initial exhaustion of the masseter muscle (determined by electromyography). The groups will then be submitted to the interventions and MVC will be performed a second time to record the time until initial exhaustion of the masseter muscle (determined by electromyography). During the procedures, the volunteers will receive verbal encouragement as well as visual feedback on the monitor to maintain MVC. Before the readings, the volunteers will undergo training of the procedure for the acquisition of the EMG signal.

CONTACTS AND LOCATIONS:
Locations (1):
- University Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No